CLINICAL TRIAL: NCT04882930
Title: Reproducibility of fNIRS Parameters During Walking in Stroke Patients and Healthy Subjects
Brief Title: Reproducibility of fNIRS Parameters During Walking
Acronym: REPROXY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Régional d'Orléans (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CHRO-2020-23
Record Dates: First submitted 2021-04-15; First posted 2021-05-12 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-08

CONDITIONS: Stroke
Keywords: fNIRS; reproductibility; stroke; gait
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Healthy subjects, acute stroke patients, subacute stroke patients
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Functional Near-Infrared Spectroscopy (fNIRS) acquisitions (Experimental): The hemodynamic response in CPF will be measured using an Octomon+ system (Artinis). Eight emission and two detector probes will be arranged on the participant's forehead.
  Interventions: Procedure: Functional Near-Infrared Spectroscopy (fNIRS)

INTERVENTIONS:
Procedure: Functional Near-Infrared Spectroscopy (fNIRS) — All participants will undergo Functional Near-Infrared Spectroscopy (fNIRS). The hemodynamic response in CPF will be measured using an Octomon+ system (Artinis). Eight emission and two detector probes will be arranged on the participant's forehead.

SUMMARY:
Brain activation can be studied using the Functional Near InfraRed Spectroscopy (fNIRS). It was shown that CPF activation during walking and during dual task could be different in stroke patients and in healthy subjects.

To date, fNIRS reliability is not completely established during walking and during dual task. Therefore, this study will examine the reproducibility of fNIRS parameters during simple walking and during dual task in healthy subjects and in stroke patients.

DETAILED DESCRIPTION:
A fNIRS system will be used to measure the CPF activation. The subjects will walk at their preferred speed on 10 m 3 times and while doing a cognitive task (dual task) 3 times also (in a random order). The same test will be repeated five minutes later. The fNIRS system will be retired and the same test will be repeated 10 min later.

ELIGIBILITY:
Inclusion Criteria:

* Acute stroke group, subacute stroke group, and control group:

  * Age 50 to 80 years
  * Affiliated with a social security plan
  * Able to walk 20 meters unassisted
* Acute Stroke and Subacute Stroke Group:

  * Stroke onset less than 14 days (for the acute stroke group) or between 14 days and 6 months (for the subacute stroke group)
  * Stroke located in the left or right middle cerebral artery.

Exclusion Criteria:

* Acute stroke group, subacute stroke group, and control group:

  * Person under guardianship or curatorship
  * Refusal to sign informed consent
  * Known rheumatologic or cardiologic history
  * Medication that alters the vigilance and may affect walking (high dose psychotropic drugs, antispastic drugs).
* Acute stroke group and subacute stroke group:

  * History of symptomatic stroke
  * Previous neurological disease limiting gait, aphasia or impaired cognitive function (mild cognitive dementia, Alzheimer's or Parkinson's disease)
  * Ambulatory functional category < 3
* Control group: neurological medical history

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2021-06-29 (Actual); Primary Completion 2023-09-08 (Actual); Study Completion 2023-09-08 (Actual)

PRIMARY OUTCOMES:
Oxyhemoglobin (HbO) variations during simple walking and during dual task | Day 0
  HbO will be measured by the NIR spectrometry technique continuously at rest and during walking. This technique allows to measure the variations of HbO concentration by measuring the variations of light absorption by the explored tissues.
Deoxyhemoglobin (HbR) variations during simple walking and during dual task | Day 0
  HbR will be measured by the NIR spectrometry technique continuously at rest and during walking. This technique allows to measure the variations of HbR concentration by measuring the variations of light absorption by the explored tissues.

SECONDARY OUTCOMES:
Oxyhemoglobin (HbO) variations of acute stroke patients | Day 0
Deoxyhemoglobin (HbR) variations of acute stroke patients | Day 0
Oxyhemoglobin (HbO) variations of subacute stroke patients | Day 0
Deoxyhemoglobin (HbR) variations of subacute stroke patients | Day 0
Oxyhemoglobin (HbO) variations using different mathematical treatments. | Day 0
Deoxyhemoglobin (HbR) variations using different mathematical treatments. | Day 0

CONTACTS AND LOCATIONS:
Overall Officials: Andreea AIGNATOAIE, Principal Investigator — CHR d'Orléans
Locations (3):
- France (3):
  - Centre de Réadaptation Fonctionnelle et d'Appareillage Le Coteau, La Chapelle-Saint-Mesmin
  - Chu Limoges, Limoges
  - CHR Orléans, Orléans

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hermand E, Tapie B, Dupuy O, Fraser S, Compagnat M, Salle JY, Daviet JC, Perrochon A. Prefrontal Cortex Activation During Dual Task With Increasing Cognitive Load in Subacute Stroke Patients: A Pilot Study. Front Aging Neurosci. 2019 Jul 2;11:160. doi: 10.3389/fnagi.2019.00160. eCollection 2019. PMID 31312136
- [Background] Hawkins KA, Fox EJ, Daly JJ, Rose DK, Christou EA, McGuirk TE, Otzel DM, Butera KA, Chatterjee SA, Clark DJ. Prefrontal over-activation during walking in people with mobility deficits: Interpretation and functional implications. Hum Mov Sci. 2018 Jun;59:46-55. doi: 10.1016/j.humov.2018.03.010. Epub 2018 Mar 29. PMID 29604488
- [Background] Holden MK, Gill KM, Magliozzi MR, Nathan J, Piehl-Baker L. Clinical gait assessment in the neurologically impaired. Reliability and meaningfulness. Phys Ther. 1984 Jan;64(1):35-40. doi: 10.1093/ptj/64.1.35. PMID 6691052
- [Background] Pelicioni PHS, Tijsma M, Lord SR, Menant J. Prefrontal cortical activation measured by fNIRS during walking: effects of age, disease and secondary task. PeerJ. 2019 May 3;7:e6833. doi: 10.7717/peerj.6833. eCollection 2019. PMID 31110922